CLINICAL TRIAL: NCT05190939
Title: The Use of Dye-less Cystoscopy in Assessing Urinary Tract Integrity During Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Eav Lim, Site Director, Gynecology Oncology, WellSpan Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1236245-7
Record Dates: First submitted 2021-12-09; First posted 2022-01-13 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Hysterectomy; Cystoscopy
Keywords: hysterectomy; universal cystoscopy; cystoscopy
MeSH Terms: interventions — Drinking Water

STUDY DESIGN:
Intervention Model Description: Patients undergoing hysterectomy are randomized to one of 4 study arms for cystoscopy: 1) dye/saline 2) dye/water 3) no-dye/saline and 4) no-dye/water
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- no-dye/saline (Active Comparator): Subjects assigned to the no-dye/saline group will have cystoscopy performed using saline as the bladder distending media and will not utilize any intravenous dye
  Interventions: Diagnostic Test: No intervention
- dye/saline (Experimental): Subjects assigned to the dye/saline group will have cystoscopy performed using saline as the bladder distending media and will utilize intravenous dye (methylene blue or fluorescein) as a ureteral jet visualization aid
  Interventions: Diagnostic Test: intravenous dye
- no-dye/water (Experimental): Subjects assigned to the no-dye/water group will have cystoscopy performed using water as the bladder distending media and will not utilize any intravenous dye
  Interventions: Diagnostic Test: water as bladder distending media
- dye/water (Experimental): Subjects assigned to the dye/water group will have cystoscopy performed using water as the bladder distending media and will utilize intravenous dye (methylene blue or fluorescein) as a ureteral jet visualization aid
  Interventions: Diagnostic Test: water as bladder distending media; Diagnostic Test: intravenous dye

INTERVENTIONS:
Diagnostic Test: water as bladder distending media — water will be used for bladder dissension during cystoscopy
  Arms: dye/water; no-dye/water
Diagnostic Test: intravenous dye — intravenous dye using methylene blue or fluorescein will be used for visual aid of ureteral jets during cystoscopy
  Arms: dye/saline; dye/water
Diagnostic Test: No intervention — Saline only, no dye
  Arms: no-dye/saline

SUMMARY:
An investigation comparing the reliability of dye-aided versus dye-less evaluation of urinary tract integrity during intra-operative cystoscopy among patients undergoing hysterectomy.

DETAILED DESCRIPTION:
Surgical injury to the urinary bladder and ureters is a recognized hazard with gynecologic procedures. Overall incidence is low; however, undetected injury to the bladder or ureter can be associated with avoidable morbidity. Approximately 75 to 85% of ureteral injuries are detected postoperatively. Various techniques have been investigated to prevent or detect genitourinary tract injuries during gynecologic surgery. Cystoscopy has been shown to increase the detection rate of urinary tract injury during gynecologic procedures compared to visual detection.

Intra-operative detection of urinary tract injury enables primary repair with high rates of success and avoidance of morbidity. Currently however, there is no standard recommendation for the routine use of cystoscopy in general gynecologic surgeries or in patients undergoing hysterectomy for gynecologic malignancies. Cost appears to be the main reason for the lack of a policy level endorsement of routine cystoscopy. One analysis concluded that ureteral injury rate was too low to justify routine cystoscopy, however other studies have reported higher urinary tract injury rates than previously published data, noted especially with the increasing use minimally invasive surgery.

Removal of dye usage with cystoscopy can help mitigate the issue of cost associated with routine cystoscopy. Various dye agents are used to aid in the visualization of urine efflux. Multiple studies have evaluated the pros and cons of these dyes. The ability to perform cystoscopy without dye would decrease cost, if the accuracy of urinary tract injury identification is not compromised. The primary objective of this study is to assess the accuracy of dye-less cystoscopy in the detection of urinary tract injury following hysterectomy. The investigators hypothesize that accurate cystoscopic evaluation for urinary tract injury at hysterectomy can be accomplished without the use of dye.

This study is a randomized prospective evaluation in which patients undergoing hysterectomy for both benign and malignant conditions are randomized into one of four study arms: 1) dye/saline 2) dye/water 3) no-dye/saline and 4) no-dye/water. Following completion of hysterectomy patients undergo routine cystoscopy utilizing distending media and dye (or no dye) according to their assigned randomization. Two independent and blinded evaluations of the bilateral ureteral jet strengths is then performed using a continuous visual scale scoring system. Ureteral jet strength scores are then evaluated for inter-observer correlation as well as comparison of jet strength and time until initial ureteral jetting is seen between the four randomized arms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 18 years of age and less than 90 years of age able to give informed consent
* Subjects undergoing hysterectomy for benign or malignant indications

Exclusion Criteria:

* Pregnancy or planned fertility
* Inability to provide informed consent
* Subject is not a surgical candidate

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients undergoing hysterectomy
Enrollment: 276 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2019-12-29 (Actual)

PRIMARY OUTCOMES:
Inter-observer correlation of urine efflux strength during cystoscopy | at time of cystoscopy
  Observers visually assess ureters on-screen simultaneously and independently. Ureteral jet efflux from each ureter is assigned a score on a linear visual scale from 0 to 5. The best of three scores of three consecutive jets from each ureter is assigned as the strength of ureteral jet. On a continuous visual scale, absent efflux is assigned as zero, slow or impaired efflux is assigned up to a score of 2, average flow neither sluggish nor brisk is assigned at least 2, and brisk flow is assigned a score of at least 3 and up to a score of 5. Evaluators determine if efflux is greater than 2. If so, evaluators are instructed to determine if efflux is 3 or 5- jets scored as 3 represent regular stream flow with no intermittent breaks and jets scored as 5 represented continuous strong flow. A score of 4 is given if the urine jet flow did not meet the criteria for a scoring of 3 or 5. Correlation of score agreement between observers and group assignments is then determined.

SECONDARY OUTCOMES:
Comparison of ureteral jet strength between groups based group assignment | at time of cystoscopy
  At time of cystoscopy ureteral jet strength is compared between the group assignments based on distending media and dye or no dye. Ureteral jet strength is measured using a continuous visual scale as with the primary outcome however the outcome focus is absolute ureteral jet strength rather than inter-observer correlation of jet strength.
Ureteral jet time | at time of cystoscopy
  Time until initial ureteral jet is observed between groups based on dye use distending media

CONTACTS AND LOCATIONS:
Overall Officials: Okechukwu Ibeanu, MD, Principal Investigator — WellSpan Health
Locations (1):
- Wellspan Health, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibeanu OA, Chesson RR, Echols KT, Nieves M, Busangu F, Nolan TE. Urinary tract injury during hysterectomy based on universal cystoscopy. Obstet Gynecol. 2009 Jan;113(1):6-10. doi: 10.1097/AOG.0b013e31818f6219. PMID 19104353
- [Background] Dowling RA, Corriere JN Jr, Sandler CM. Iatrogenic ureteral injury. J Urol. 1986 May;135(5):912-5. doi: 10.1016/s0022-5347(17)45921-0. PMID 3959239
- [Background] Chou MT, Wang CJ, Lien RC. Prophylactic ureteral catheterization in gynecologic surgery: a 12-year randomized trial in a community hospital. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jun;20(6):689-93. doi: 10.1007/s00192-008-0788-3. Epub 2009 Jan 23. PMID 19165412
- [Background] Redan JA, McCarus SD. Protect the ureters. JSLS. 2009 Apr-Jun;13(2):139-41. PMID 19660205
- [Background] Frankel J. Accuracy of cystoscopy in the diagnosis of ureteral injury in benign gynecologic surgery. Int Urogynecol J Pelvic Floor Dysfunct. 2004 Mar-Apr;15(2):75. doi: 10.1007/s00192-004-1144-x. Epub 2004 Feb 20. No abstract available. PMID 15014932
- [Background] Gilmour DT, Das S, Flowerdew G. Rates of urinary tract injury from gynecologic surgery and the role of intraoperative cystoscopy. Obstet Gynecol. 2006 Jun;107(6):1366-72. doi: 10.1097/01.AOG.0000220500.83528.6e. PMID 16738165
- [Background] Teeluckdharry B, Gilmour D, Flowerdew G. Urinary Tract Injury at Benign Gynecologic Surgery and the Role of Cystoscopy: A Systematic Review and Meta-analysis. Obstet Gynecol. 2015 Dec;126(6):1161-1169. doi: 10.1097/AOG.0000000000001096. PMID 26551173
- [Background] Barber EL, Polan RM, Strohl AE, Siedhoff MT, Clarke-Pearson DL. Cystoscopy at the Time of Hysterectomy for Benign Indications and Delayed Lower Genitourinary Tract Injury. Obstet Gynecol. 2019 May;133(5):888-895. doi: 10.1097/AOG.0000000000003192. PMID 30969213
- [Background] American College of Obstetricians and Gynecologists. ACOG Committee Opinion. Number 372. July 2007. The Role of cystourethroscopy in the generalist obstetrician-gynecologist practice. Obstet Gynecol. 2007 Jul;110(1):221-224. doi: 10.1097/01.AOG.0000263916.77694.20. PMID 17601926
- [Background] Visco AG, Taber KH, Weidner AC, Barber MD, Myers ER. Cost-effectiveness of universal cystoscopy to identify ureteral injury at hysterectomy. Obstet Gynecol. 2001 May;97(5 Pt 1):685-92. doi: 10.1016/s0029-7844(01)01193-0. PMID 11339916
- [Background] Vakili B, Chesson RR, Kyle BL, Shobeiri SA, Echols KT, Gist R, Zheng YT, Nolan TE. The incidence of urinary tract injury during hysterectomy: a prospective analysis based on universal cystoscopy. Am J Obstet Gynecol. 2005 May;192(5):1599-604. doi: 10.1016/j.ajog.2004.11.016. PMID 15902164
- [Background] Espaillat-Rijo L, Siff L, Alas AN, Chadi SA, Zimberg S, Vaish S, Davila GW, Barber M, Hurtado EA. Intraoperative Cystoscopic Evaluation of Ureteral Patency: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1378-1383. doi: 10.1097/AOG.0000000000001750. PMID 27824741
- [Background] Siff LN, Unger CA, Jelovsek JE, Paraiso MF, Ridgeway BM, Barber MD. Assessing ureteral patency using 10% dextrose cystoscopy fluid: evaluation of urinary tract infection rates. Am J Obstet Gynecol. 2016 Jul;215(1):74.e1-6. doi: 10.1016/j.ajog.2016.02.006. Epub 2016 Feb 12. PMID 26875949
- [Background] Grimes CL, Patankar S, Ryntz T, Philip N, Simpson K, Truong M, Young C, Advincula A, Madueke-Laveaux OS, Walters R, Ananth CV, Kim JH. Evaluating ureteral patency in the post-indigo carmine era: a randomized controlled trial. Am J Obstet Gynecol. 2017 Nov;217(5):601.e1-601.e10. doi: 10.1016/j.ajog.2017.07.012. Epub 2017 Jul 18. PMID 28729014
- [Background] Propst K, Tunitsky-Bitton E, O'Sullivan DM, Steinberg AC, LaSala C. Phenazopyridine for Evaluation of Ureteral Patency: A Randomized Controlled Trial. Obstet Gynecol. 2016 Aug;128(2):348-355. doi: 10.1097/AOG.0000000000001472. PMID 27399998
- [Background] Strom EM, Chaudhry ZQ, Guo R, Maisonet AJ, Holschneider CH, Wieslander CK. Effectiveness of Assessing Ureteral Patency Using Preoperative Phenazopyridine. Female Pelvic Med Reconstr Surg. 2019 Jul/Aug;25(4):289-293. doi: 10.1097/SPV.0000000000000540. PMID 29300258
- [Background] Hui JYC, Harvey MA, Johnston SL. Confirmation of ureteric patency during cystoscopy using phenazopyridine HCl: a low-cost approach. J Obstet Gynaecol Can. 2009 Sep;31(9):845-849. doi: 10.1016/S1701-2163(16)34303-1. PMID 19941709
- [Background] Cohen SA, Chaudhry Z, Oliver JL, Kreydin EI, Nguyen MT, Mills SA, Ackerman AL, Kim JH, Tarnay CM, Raz S. Comparison of Times to Ureteral Efflux after Administration of Sodium Fluorescein and Phenazopyridine. J Urol. 2017 Feb;197(2):519-523. doi: 10.1016/j.juro.2016.07.099. Epub 2016 Sep 21. PMID 27664579